CLINICAL TRIAL: NCT03047889
Title: A Nation-wide Multicenter Clinical Epidemiologic Study of Chinese Females With Advanced Breast
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Binghe Xu, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CH-BC-045
Record Dates: First submitted 2016-11-29; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: standard therapy — standard therapy for advanced/metastatic breast cancer

SUMMARY:
To study the epidemiological trends and characteristics for advanced breast cancer patients, to analyze these trends and report the results

DETAILED DESCRIPTION:
In this study, the investigators conducted a hospital-based retrospective clinical study, recruiting female advanced breast cancer patients from 14 tertiary hospitals at 7 classic geographic regions, to study the clinical epidemiologic characteristics of advanced breast cancer and the current standard of clinical diagnosis and treatment in order to provide references for standardized treatment therapy, and to improve the quality of life and prolong survival time.

To study the epidemiological trends and characteristics for advanced BC patients, to analyze these trends and report the results. To learn about the current treatment therapy for advanced BC patients in different areas in China.To provide references for standardized treatment therapy, to improve the quality of patients' life and to prolong the survival time for the advanced BC patients.To assess the different treatment therapies for advanced BC with consideration of economic cost-effectiveness

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as advanced breast cancer during Jan1st,2012-Dec31st,2014
* complete with surgical pathology data, auxiliary treatment, there is a clear recurrence, transfer time, place, transfer of recurrence after treatment, and curative effect evaluation details.In any age, ethnic group cases.

Exclusion Criteria:

* no available medical record

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 21 hospitals were selected in this study. The investigators recruited 4200 advanced BC cases, who were first diagnosed with advanced BC from January 1st, 2012 to December 31st, 2014 from these hospitals.
Sampling Method: Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Survival status at 3 years | 3 years
  percentage of patients still alive at 3 years

SECONDARY OUTCOMES:
PFS | 3 years
  Progression-free survival of first line therapy
Survival status at 5 years | 3 years
  percentage of patients still alive at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Principal Investigator — Chinese Academy of Medical Sciences; Youlin Qiao, Principal Investigator — Chinese Academy of Medical Sciences
Locations (19):
- China (19):
  - The 307th Hospital of Military Medical Sciences, Beijing
  - Sichuan Cancer Hospital and Institute, Chengdu
  - The First Affliated Hospital of Chongqing Medical University, Chongqing
  - FuZhou General Hospital of National Miltary Command, Fuzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Henan Cancer Hospital, Henan
  - Hunan Cancer Hospital, Hunan
  - Jiangsu Provinces hospital, Jiangsu
  - Tumor Hospital of Yunnan Province, Kunming
  - Liaoning Cancer Hospital, Zhejiang Cancer Hospital, Liaoning
  - General Hospital of NingXia Medical University, Ningxia
  - Fudan University Shanghai Cancer Center, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - The First Hospital of Xi'an Jiaotong University, Xi'an
  - Xinjiang Medical University Cancer Hospital, Xinjiang
  - FuJian Provincial Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han YQ, Yi ZB, Yu P, Wang WN, Ouyang QC, Yan M, Wang XJ, Hu XC, Jiang ZF, Huang T, Tong ZS, Wang SS, Yin YM, Li H, Yang RX, Yang HW, Teng YE, Sun T, Cai L, Li HY, Ouyang XN, He JJ, Liu XL, Yang SE, Qiao YL, Fan JH, Wang JY, Xu BH. Comparisons of Treatment for HER2-Positive Breast Cancer between Chinese and International Practice: A Nationwide Multicenter Epidemiological Study from China. J Oncol. 2021 Sep 15;2021:6621722. doi: 10.1155/2021/6621722. eCollection 2021. PMID 34567118
- [Derived] Guo F, Yi Z, Wang W, Han Y, Yu P, Zhang S, Ouyang Q, Yan M, Wang X, Hu X, Jiang Z, Huang T, Tong Z, Wang S, Yin Y, Li H, Yang R, Yang H, Teng Y, Sun T, Cai L, Li H, Chen X, He J, Liu X, Yang S, Fan J, Qiao Y, Wang J, Xu B. Profile, treatment patterns, and influencing factors of anthracycline use in breast cancer patients in China: A nation-wide multicenter study. Cancer Med. 2021 Oct;10(19):6744-6761. doi: 10.1002/cam4.4215. Epub 2021 Sep 2. PMID 34472719
- [Derived] Wu Y, Han Y, Yu P, Ouyang Q, Yan M, Wang X, Hu X, Jiang Z, Huang T, Tong Z, Wang S, Yin Y, Li H, Yang R, Yang H, Teng Y, Sun T, Cai L, Li H, Chen X, He J, Liu X, Yang S, Qiao Y, Fan J, Wang J, Xu B. Endocrine Therapy for Hormone Receptor-Positive Advanced Breast Cancer: A Nation-Wide Multicenter Epidemiological Study in China. Front Oncol. 2021 Feb 11;10:599604. doi: 10.3389/fonc.2020.599604. eCollection 2020. PMID 33643905
- [Derived] Yi ZB, Yu P, Zhang S, Wang WN, Han YQ, Ouyang QC, Yan M, Wang XJ, Hu XC, Jiang ZF, Huang T, Tong ZS, Wang SS, Yin YM, Li H, Yang RX, Yang HW, Teng YE, Sun T, Cai L, Li HY, Chen X, He JJ, Liu XL, Yang SE, Wang JY, Fan JH, Qiao YL, Xu BH. Profile and outcome of receptor conversion in breast cancer metastases: a nation-wide multicenter epidemiological study. Int J Cancer. 2021 Feb 1;148(3):692-701. doi: 10.1002/ijc.33227. Epub 2020 Aug 19. PMID 32700765